CLINICAL TRIAL: NCT01046695
Title: Evaluating Efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) for Postoperative Pain After Video-Assisted Thoracotomy Surgery (VATS)
Brief Title: Evaluating Transcutaneous Electrical Nerve Stimulation for Postoperative Pain After Video-Assisted Thoracotomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deborah Engen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-000141
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Postoperative Pain
Keywords: VATS; Video-Assisted Thoracotomy; Thoracic Surgery, Video-Assisted
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS Unit (Active Comparator): This arm will be adding the use of the TENS unit for 48 hours in addition to standard care for their post operative pain control.
  Patient's primary area of postoperative pain was determined by nursing personnel. Four electrodes were placed on or around the area of maximum pain. The TENS unit was turned on, 1 of 5 frequency patterns selected and the impulse turned up until the patient could feel the impulse. The location of the electrodes, the pattern, and/or the intensity of the TENS unit were adjusted until the patient achieved maximum comfort with the sensation.
  Interventions: Device: TENS Unit
- Control Arm (No Intervention): This arm will have standard care for their post operative pain control.

INTERVENTIONS:
Device: TENS Unit — TENS is a method of pain relief that uses a battery operated electronic device with cutaneously applied electrodes that deliver electrical signals to peripheral nerves through the intact skin. The TENS Unit is a low voltage system that will only be used to a level to create alternative to pain sensation and will not create muscle response.
  Other Names: Transcutaneous Electrical Nerve Stimulation unit
  Arms: TENS Unit

SUMMARY:
We propose to evaluate the use of Transcutaneous Electrical Nerve Stimulation (TENS) in patients having undergone Video-Assisted Thoracotomy Surgery (VATS) with the aim to determine if:

* Nurses will be able to apply TENS effectively and in a timely manner to post VATS patients.
* Use of TENS immediately after thoracic surgery and for the first 48 hours will add to patient's pain control.
* Tens will reduce medication use.
* Tens will reduce nausea and vomiting.

DETAILED DESCRIPTION:
Video-Assisted Thoracotomy (VATS) patient's post procedure pain is a significant problem that may delay the recovery of thoracic surgery patients. Without adequate control of pain, the patient's mobilization and ability to participate in bronchial hygiene is compromised increasing the risk for pulmonary complications and inhibiting the body's natural healing ability. When acute post VATS pain is poorly controlled, the incidence of chronic post VATS pain six months or longer after the surgery increases. Post-operative pain is controlled largely through the use of pain medications delivered by a variety of routes including: epidural, intravenous, and when able, oral. Medications used include opioids which have side effects such as nausea, dizziness, drowsiness and constipation that may further delay the patient's recovery and prolong the hospital stay.

Transcutaneous Electrical Nerve Stimulation (TENS) is a method of pain relief that uses cutaneously applied electrodes that deliver electrical signals to peripheral nerves through the intact skin. Treating pain with TENS results in the patient having a reduced perception of pain. The effectiveness of TENS is based on two mechanisms: 1) the gate control theory of pain relief where stimulation of myelinated sensory fibers disrupts neuronal processing in the substantia gelatinosa of the spinal cord, and 2) the stimulation-induced release of endogenous opioids, both in the central nervous system and the general circulation. The present practice for obtaining and applying a TENS unit on a patient for pain relief requires consultation with Physical Therapy who will come and assess the patient and then apply the TENS unit and make recommendations for settings and therapy. This process limits the response to only daytime and often results in a delay in initiation of treatment. After providing education and training it is anticipated that nurses could successfully apply a TENS unit and initiate therapy early in the immediate post operative period. The more timely application of a TENS unit to a post VATS patient could improve pain management outcomes for this population.

Patient's primary area of postoperative pain was determined by nursing personnel. Four electrodes were placed on or around the area of maximum pain by nurses trained in TENS therapy. The TENS unit was turned on, 1 of 5 frequency patterns selected and the impulse turned up until the patient could feel the impulse. The 5 program options available included: #1. Alternate Ramped Burst (ARB) (Rate = 100 pps; Ramp Up Time = 0.5s; On Time = 5s; Off Time = 6s). #2. Simple Modulated Pulse (SMP) (Rate = 125 pps; Cycle Time = 12s; Span Percentage = 40%; Rate stays in the 2-10 pps range for 1/3 of the cycle time (4 seconds) as the rate modulates down to 2 pulses per second (pps) and then back up again. #3. Modulated Amplitude (MA) (Rate = 125 pps; Cycle Time = 1s; Span Percentage = 60%). #4. Simple Modulated Pulse (SMP) (Rate = 125 pps; Cycle Time = 12s; Span Percentage = 40%; Rate stays in the 2-10 pps range for 1/3 of the cycle time (4 seconds) as the rate modulates down to 2 pulses per second (pps) and then back up again). #5 Modulated Amplitude, MA (Rate = 125 pps; Cycle Time = 1s; Span Percentage = 60%). The location of the electrodes, the pattern, and/or the intensity of the TENS unit were adjusted until the patient achieved maximum comfort with the sensation. Five minutes after initiation of TENS therapy and every hour there after - while patient was awake- for a total of 48 hours, the patient was reassessed by nursing staff and TENS settings were adjusted for patient comfort and pain control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-100 able to give informed consent.
* Able to speak and understand English.

Exclusion Criteria:

* Too confused to provide data or not extubated within 48 hours after surgery.
* Unable to speak and understand English.
* Patients with active internal pacer wires, demand type implanted pacemakers or defibrillator.
* Transplant patients.
* Children, prisoners, any woman who is pregnant.
* Patients that are non-scheduled surgery cases or occurring Saturday or Sunday.
* Ventricular Assisted Device (VAD) patients.
* Know allergies or intolerance to TENS electrodes.
* Patients who have had the Da Vinci robotic assisted minimally invasive procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Engen, O.T., Principal Investigator — Mayo Clinic; Dietlind L. Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Engen DJ, Carns PE, Allen MS, Bauer BA, Loehrer LL, Cha SS, Chartrand CM, Eggler EJ, Cutshall SM, Wahner-Roedler DL. Evaluating efficacy and feasibility of transcutaneous electrical nerve stimulation for postoperative pain after video-assisted thoracoscopic surgery: A randomized pilot trial. Complement Ther Clin Pract. 2016 May;23:141-8. doi: 10.1016/j.ctcp.2015.04.002. Epub 2015 Apr 20. PMID 25935320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from individuals undergoing video-assisted thoracic surgery at the Mayo Clinic in Rochester, Minnesota from March 18 through September 22, 2010.
Pre-assignment Details: 56 subjects enrolled, but 14 subjects didn't start and receive the intervention. On the TENS Unit arm, 1 went straight to the ICU, 1 refused stating "no pain to treat", and 4 did not have a VATS or had a thoracotomy. On the control arm, 1 did not have a VATS, 1 had an defibrillator, 3 went straight to the ICU, and 3 did not get started by nursing.
Groups:
- Control Arm: Once awake from surgery this arm had standard care for 48 hours for their postoperative pain control using each surgeons usual postoperative medications and procedures.
- TENS Unit: Once awake from surgery this arm added the use of the TENS unit for 48 hours in addition to standard care for their postoperative pain control. The TENS unit was set to each patients individual preference which included intensity, frequency and the placement of where they wanted the electrodes.
Period: Overall Study
Arm/Group | Control Arm | TENS Unit
Started | 20 | 22
Completed | 20 | 20
Not Completed | 0 | 2
Not completed — Subject had a pacemaker | 0 | 1
Not completed — TENS interfered with the cardiac monitor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TENS Unit | Control Arm | Total
Number analyzed (Participants) | 22 | 20 | 42
Age Continuous [Median (Full Range); unit: years] | 63 [30 to 78] | 63 [41 to 84] | 63 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Secondary Outcome: Mean Opioid Use, Converted Into Oral Morphine Equivalents (OME) at 24 and 48 Hours
Description: As subjects could have been prescribed many different analgesics, the amount of pain medication was converted to the standard oral morphine equivalents (OME), so that the mean dose needed could be compared.
Time Frame: 24 hours and 48 hours after awakening from video-assisted thoracic surgery
Measure: Mean (Standard Deviation); unit: mg of oral morphine
Arm/Group | TENS Unit | Control Arm
Number analyzed (Participants) | 20 | 20
mg of oral morphine
  24 hours | 90.19 (48.08) | 93.65 (89.65)
  48 hours | 47.50 (55.67) | 69.68 (113.65)
Statistical Analysis 1: Comparison: TENS Unit; Decrease in OME use in the TENS Unit during the first and second 24 hours; Test type: Superiority or Other; p = .005, t-test, 2 sided
Statistical Analysis 2: Comparison: Control Arm; Decrease in OME use in the Control Arm during the first and second 24 hours; Test type: Superiority or Other; p = .11, t-test, 2 sided

2. Secondary Outcome: Satisfaction With Pain Control at 48 Hours
Description: Pain control was measured by using a Visual Analog Scale (VAS) with a range from 0-10; with 0 being very satisfied and 10 being very dissatisfied.
Time Frame: 48 hours after awakening from video-assisted thoracic surgery
Population: 11 participants on each arm did not complete the VAS.
Measure: Number; unit: participants
Arm/Group | TENS Unit | Control Arm
Number analyzed (Participants) | 20 | 20
participants
  Satisfaction Score 0 (very satisfied) | 2 | 2
  Satisfaction Score 1 | 1 | 2
  Satisfaction Score 2 | 0 | 2
  Satisfaction Score 3 | 1 | 1
  Satisfaction Score 4 | 2 | 0
  Satisfaction Score 5 | 1 | 1
  Satisfaction Score 6 | 1 | 0
  Satisfaction Score 7 | 0 | 0
  Satisfaction Score 8 | 0 | 0
  Satisfaction Score 9 | 1 | 1
  Satisfaction Score 10 | 0 | 0
  Unknown | 11 | 11
Statistical Analysis 1: Comparison: TENS Unit vs Control Arm; Test type: Superiority or Other; p = .70, t-test, 2 sided

3. Primary Outcome: Mean Pain Score
Description: Pain was measured by using the Visual Analog Scale (VAS) with a range from 1-10; with 0 being no pain and 10 being severe pain. Pain scores were measured from hour 1 to hour 48 for each patient. Some scores were missed when patients were asleep. In these cases, the previous score was used.
Time Frame: hour 1 to hour 48 after awakening from video-assisted thoracic surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TENS Unit | Control Arm
Number analyzed (Participants) | 20 | 20
units on a scale
  Hour 1 | 4.55 (3.02) | 3.85 (2.39)
  Hour 2 | 4.30 (3.28) | 3.80 (2.09)
  Hour 3 | 4.30 (2.94) | 3.95 (1.73)
  Hour 4 | 3.55 (3.05) | 4.25 (1.59)
  Hour 5 | 2.90 (2.43) | 3.80 (1.51)
  Hour 6 | 2.75 (2.20) | 3.45 (1.99)
  Hour 7 | 2.80 (2.17) | 3.60 (2.16)
  Hour 8 | 3.10 (2.38) | 4.0 (1.86)
  Hour 9 | 3.05 (2.42) | 4.20 (2.09)
  Hour 10 | 2.95 (2.24) | 3.45 (2.09)
  Hour 11 | 3.25 (2.40) | 3.55 (2.11)
  Hour 12 | 3.85 (3.03) | 4.05 (2.54)
  Hour 13 | 3.50 (2.61) | 3.85 (2.60)
  Hour 14 | 3.85 (2.32) | 2.90 (1.92)
  Hour 15 | 3.55 (2.21) | 2.60 (1.98)
  Hour 16 | 3.55 (2.40) | 2.80 (2.07)
  Hour 17 | 2.70 (1.75) | 2.90 (1.62)
  Hour 18 | 2.95 (2.06) | 3.05 (1.54)
  Hour 19 | 2.95 (2.01) | 2.50 (1.67)
  Hour 20 | 3.15 (2.25) | 2.55 (1.36)
  Hour 21 | 3.20 (2.29) | 3.05 (2.11)
  Hour 22 | 3.10 (2.32) | 2.70 (1.81)
  Hour 23 | 2.75 (2.05) | 2.45 (1.67)
  Hour 24 | 2.95 (1.88) | 2.45 (1.91)
  Hour 25 | 2.50 (1.73) | 2.45 (1.82)
  Hour 26 | 2.85 (1.84) | 2.45 (1.82)
  Hour 27 | 2.65 (1.50) | 2.40 (1.98)
  Hour 28 | 2.35 (1.87) | 2.60 (2.14)
  Hour 29 | 2.60 (1.98) | 2.70 (1.84)
  Hour 30 | 1.95 (1.79) | 2.40 (1.96)
  Hour 31 | 2.10 (1.86) | 2.45 (1.93)
  Hour 32 | 2.00 (1.78) | 2.30 (1.92)
  Hour 33 | 2.05 (2.04) | 2.20 (2.14)
  Hour 34 | 2.20 (1.88) | 2.35 (2.23)
  Hour 35 | 2.10 (1.86) | 2.00 (1.92)
  Hour 36 | 2.45 (2.76) | 2.10 (2.5)
  Hour 37 | 2.80 (2.73) | 2.60 (2.33)
  Hour 38 | 2.75 (2.73) | 2.45 (2.04)
  Hour 39 | 2.50 (2.28) | 2.45 (2.14)
  Hour 40 | 2.50 (2.21) | 2.55 (1.96)
  Hour 41 | 2.30 (2.11) | 2.50 (2.01)
  Hour 42 | 1.85 (1.31) | 2.50 (2.31)
  Hour 43 | 1.70 (1.42) | 2.65 (2.30)
  Hour 44 | 1.95 (1.54) | 2.70 (2.16)
  Hour 45 | 1.70 (1.49) | 2.55 (2.09)
  Hour 46 | 1.75 (1.52) | 2.50 (1.93)
  Hour 47 | 1.85 (1.66) | 2.40 (2.01)
  Hour 48 | 1.75 (1.68) | 2.35 (2.23)

ADVERSE EVENTS:
Time Frame: Subjects were followed for adverse events for 48 hours after the video-assisted thoracotomy surgery.
Arm/Group | TENS Unit | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 1/22 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TENS Unit (N=22) | Control Arm (N=20)
TENS interfered with cardiac monitor (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes